CLINICAL TRIAL: NCT06056180
Title: Investigation of the Effects of Motor Imagery Training Given With Action Observation on Balance Performance in Geriatric Individuals
Brief Title: The Effect of Motor Image Training on Balance Performance in Geriatric Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Şeyda Ercan Yüceer, Research Assistant, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSKUSYuceer_001
Record Dates: First submitted 2023-06-12; First posted 2023-09-28 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Imagery (Psychotherapy); Postural Control; Postural Balance; Virtual Reality Therapy; Surface Electromyography; Geriatric Assessment; Physical Therapy Techniques; Physical Therapy; Healthy Ageing; Healthy Aging; Falling
Keywords: visual motor imagery; kinesthetic motor imagery; postural control; virtual reality therapy; interactive video games; balance platform with pressure sensor; surface electromyography; balance confidence; fall risk; mobility; cognitive processing speed; smartphone gyroscope sensor dataset; action observation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The person among the researchers who will evaluate the individuals will be blinded to the treatment.
  The person who will make the statistical evaluations of the data will be blind to the treatment and evaluations to be made to the individuals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance Training+ Action Observation Training + Motor İmagery Training (Experimental): The study group (23 cases) will be given motor imagery training and virtual reality-based balance training along with action observation.
  Interventions: Other: Balance Training; Other: Motor İmagery Training; Other: Action Observation Training
- Balance Training (Active Comparator): Only virtual reality-based balance training will be given to the control group (23 cases).
  Interventions: Other: Balance Training

INTERVENTIONS:
Other: Balance Training — Participants will be given static and dynamic balance training with a balance platform game console (20 minutes) containing interactive video games based virtual reality for a total of 6 weeks.
Other: Motor İmagery Training — For motor imagery training, two visualization scenarios will be created: anterior and posterior motor imagery. One of the visualization scenarios appropriate to each individual's needs will be used. Participants will be asked to perform kinesthetic or visual motor imagery in accordance with the scenario they listened to (10 minutes).
  Arms: Balance Training+ Action Observation Training + Motor İmagery Training
Other: Action Observation Training — Action observation training will be done using video modeling method. The video content will include Nintendo Wii games in which the games that the person will play in that session are played by someone else and successful scores are achieved (10 minutes).
  Arms: Balance Training+ Action Observation Training + Motor İmagery Training

SUMMARY:
The goal of this study [type of study: clinical trial] is to was planned to investigate the effect of motor imagery training given to geriatric individuals with action observation on their balance performance and to compare these two methods.

The main questions it aims to answer are:

1. Is virtual reality-based balance training given together with action observation and motor imagery for six weeks in geriatric individuals more effective in improving static balance than virtual reality-based balance training given alone?
2. Is virtual reality-based balance training given together with action observation and motor imagery for six weeks in geriatric individuals more effective in improving dynamic balance than virtual reality-based balance training given alone?
3. Is virtual reality-based balance training given together with motor imagery for six weeks in geriatric individuals more effective in increasing balance confidence than virtual reality-based balance training given alone?

46 geriatric individuals will be randomized into 2 groups. Along with action observation, motor imagery training and virtual reality-based balance training will be given to the study group. On the other hand, only virtual reality-based balance training will be given to the control group. All assessments will be repeated before and after the trainings. The trainings will be applied 2 days a week for 6 weeks. Each training session; 25 minutes for the control group and 45 minutes for the study group.

DETAILED DESCRIPTION:
Muscle strength, proprioception, joint mobility, vestibular losses and vision losses may occur with the aging process. These losses may lead to a decrease in the ability of geriatric individuals to adapt to environmental factors. This loss of harmony may cause balance disorders in individuals by affecting static and dynamic postural control performance. Looking at the literature, balance trainings, functional exercises, flexibility, muscle strength and endurance trainings, Tai Chi, Qigong-like yoga exercises, dance, walking programs, motor imagery training given with traditional methods or virtual reality systems for the purpose of improving balance and postural control. There are studies showing the effectiveness of many methods in geriatric individuals. However, no study has been found that examines and compares the effects of virtual reality-based balance training and motor imagery training combined with action observation in addition to virtual reality-based balance training in geriatric individuals. For this reason, this study was planned to investigate the effect of motor imagery training given to geriatric individuals with action observation on their balance performance and to compare these two methods.

The study, which was designed as a prospective, randomized controlled, cross-sectional, single-blind (evaluator), will include 46 geriatric individuals aged 60 and over. The study will be initiated with individuals who meet the inclusion/exclusion criteria of the study. 46 geriatric individuals will be randomized into 2 groups. The study group (23 cases) will be given motor imagery training and virtual reality-based balance training along with action observation. Only virtual reality-based balance training will be given to the control group (23 cases). First of all, age, gender, height, body weight, upper extremity dominant side, lower extremity dominant side, body mass index, smoking history, alcohol consumption, occupation, employment status, chronic diseases, regularly used drugs, history of falling and staggering, history and pedigree information, independence in daily living activities, ability to walk 10 meters without any walking aid will be recorded. In the first evaluation before the training, the measurement of the electrical potential changes known as muscle motor unit action potentials of the subjects during the postural swings will be evaluated with the electromyography biofeedback device. Static and dynamic balance assessments will be evaluated with computerized kinesthetic balance device, Berg Balance Scale and 10 Meter Walk Test. Three-axis (x, y and z) evaluation of body oscillations will be made with an android-based smartphone application. Motor imagery skills will be evaluated with the Movement Imagination Questionnaire-3 (HIA-3) and the mental stopwatch test. All assessments will be repeated before and after the training (6 weeks later) by a researcher blinded to the training. As a training protocol, individuals in both groups will be given static and dynamic balance training with a balance platform game console (20 minutes) containing interactive video games based virtual reality for a total of 6 weeks. Before the balance training, a 5-minute relaxation training will be given to both groups. In addition to the virtual reality-based balance and relaxation training, the study group will be given motor imagery training (10 min + 10 min) with action observation before the balance training. The trainings will be applied 2 days a week for 6 weeks. Each training session; 25 min for the control group. (Relaxation training (5 min) + virtual reality-based balance training (20 min), 45 min for the study group. (Relaxation training (5 min) + motor imagery training (20 min) + virtual reality-based balance training (20 min) with action observation. All questionnaires, scales, tests and devices used in the initial evaluations will be repeated for the individuals in both groups at the end of the 6-week training. The effectiveness of the trainings will be compared with appropriate statistical methods within and between groups and discussed in the light of the literature.

ELIGIBILITY:
Inclusion Criteria:

1. To be between 60-80 years old
2. Having the ability to speak, read, understand and write Turkish
3. To have the cognitive skills to understand and apply the trainings to be applied in the study (with ≥ 24 points from the Mini Mental State Test)
4. Being able to do activities of daily living independently
5. Being able to walk independently (without using a walking aid and at least 10 meters)
6. Having a body mass index of <35 kg/m2 (not being severely obese or morbidly obese)

Exclusion Criteria:

1. Having visual, hearing and sensory impairment
2. To have had a trauma, lesion or surgery that may affect balance and musculoskeletal system in the last 6 months
3. Having a history of 2 ≥ falls in the last 6 months
4. Having any chronic lower extremity pain
5. Having an acute or chronic illness that may cause problems with balance and falling
6. Being diagnosed with sensory, vestibular and cerebellar ataxia
7. Being on any medication that may cause problems with balance, focus, attention and falling.
8. Exercising regularly, which may affect performance results
9. To stop participating in the study for any reason

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of Muscle Activities During Postural Swings | 1 day before starting treatment and First day after 6 weeks of treatment (2 times in total)
  EMG Biofeedback device will be used to evaluate the muscle activities in the lower leg anterior (m. tibialis anterior) and posterior group (m. gastrocnemius lateralis) muscles while performing postural swings.
Berg Balance Scale | 1 day before starting treatment-First day after 6 weeks of treatment (2 times in total)
  In this scale, the individual tries to maintain her balance during 14 different activities in which the center of gravity varies and is suitable for daily life activities.The total score on the Berg Balance Scale was 56. Low scores from the scale indicate a high risk of falling.
Portable computerized kinesthetic balance device of participants' static and dynamic balance | 1 day before starting treatment-First day after 6 weeks of treatment (2 times in total)
  Static and dynamic balance will be evaluated while participants stand on one or two legs on the device (eyes open/closed, in 9 different conditions). The Balance Index Score (DI) displayed on the screen as a result of the test will be recorded as the individual's balance score. The score range is 0-6000. 0 is the best score.
10 meter Walking Test | 1 day before starting treatment-First day after 6 weeks of treatment (2 times in total)
  How long it takes individuals to walk a distance of 10 meters will be recorded in seconds.
Activity-Specific Balance Confidence Scale | 1 day before starting treatment and First day after 6 weeks of treatment (2 times in total)
  The Activity-Specific Balanced Confidence Scale will be used to measure balance confidence. The total score ranges from 0 to 100, with higher scores indicating greater confidence.
Movement Imagination Questionnaire-3 | 1 day before starting treatment-First day after 6 weeks of treatment (2 times in total)
  In the questionnaire consisting of 12 items, kinesthetic, internal and external visual imagination abilities are evaluated separately.Higher scores on the survey indicate better mental imagery ability.
Mental Stopwatch Test | 1 day before starting treatment-First day after 6 weeks of treatment (2 times in total)
  Time Up and Go Test (TUG) will be used to look at the temporal similarity between the durations of real and imagined movement in geriatric individuals. Both test results will be recorded in seconds. The temporal harmony between real and imagined movement will be calculated in delta time. Higher delta time indicates lower motor imagery ability.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyda Ercan Yüceer, Principal Investigator — Mugla Sitki Kocman Univercity
Locations (1):
- Mugla Sitki Kocman University, Menteşe, Muğla, Turkey (Türkiye)